CLINICAL TRIAL: NCT04107870
Title: Efficiency of Virtual Reality Exposure Therapy in the Management of Body Dysmorphic Disorder in Female Adolescents With Anorexia Nervosa: a Randomized, Controlled Superiority Study
Brief Title: Efficiency of Virtual Reality Exposure Therapy in the Management of Body Dysmorphic Disorders in Female Adolescents With Anorexia Nervosa
Acronym: ANO-TERV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PR19054
Record Dates: First submitted 2019-09-26; First posted 2019-09-27 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Anorexia Nervosa
Keywords: ANOREXIA NERVOSA; FEMALE ADOLESCENTS; BODY DYSMORPHIC DISORDER; VIRTUAL REALITY EXPOSURE THERAPY
MeSH Terms: conditions — Anorexia Nervosa; Body Dysmorphic Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Exposure Therapy (Experimental): Female adolescents aged 13 to 18 are proposed virtual reality exposure therapy sessions, accompanied by a cognitive and behavioral therapy (CBT) therapist, to work on their body representations
  Interventions: Behavioral: Virtual Reality Exposure Therapy sessions
- Psychomotor Therapy (Active Comparator): Psychomotor therapy sessions are proposed to female adolescents aged 13 to 18 years, ac-companied by a psychomotor therapist, to work on their body representations.
  Interventions: Behavioral: Psychomotor therapy sessions

INTERVENTIONS:
Behavioral: Virtual Reality Exposure Therapy sessions — Female adolescents aged 13 to 18 are proposed virtual reality exposure therapy sessions, accompanied by a cognitive and behavioral therapy (CBT) therapist, to work on their body representations
  Arms: Virtual Reality Exposure Therapy
Behavioral: Psychomotor therapy sessions — Psychomotor therapy sessions are proposed to female adolescents aged 13 to 18 years, ac-companied by a psychomotor therapist, to work on their body representations.
  Arms: Psychomotor Therapy

SUMMARY:
Anorexia nervosa is defined in DSM V as a quantitative and qualitative dietary restriction resulting in significant weight loss, intense fear of weight gain, altered weight and body shape perception (body dysmorphic disorder) and low self-esteem influenced by weight or body shape. Body dysmorphic disorder is the most difficult symptom to manage in anorexia nervosa and its persistence is a factor associated with relapse.

Virtual reality exposure therapy has proven its effectiveness in the management of post-traumatic stress disorder in the military and is a widely used therapy. The effectiveness of this treatment using new technologies has not yet been studied for the treatment of body dysmorphic disorder in anorexia nervosa and is not used routinely. It could represent an interesting alternative to the physical approach in psychomotor therapy, traditionally offered to patients suffering from anorexia nervosa. It is important to evaluate the effectiveness of virtual reality exposure therapy in the management of body dysmorphic disorder in patients with anorexia nervosa by comparing these two care techniques.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effectiveness of Virtual Reality Exposure Therapy in the management of body dysmorphic disorder in patients with anorexia nervosa, compared to the traditionally proposed body approach in psychomotor therapy.

ELIGIBILITY:
Inclusion criteria :

* Female adolescents aged 13 to 18
* with a diagnosis of anorexia nervosa of all types (including purgative and hyperphagic) according to the DSM-V
* French as first language
* agreed to participate in the study
* parental authority holders accepting her participation in the study
* affiliated to a social security system

Patients will not be included in the study:

* with a somatic severity criterion:

  * Total aphagia
  * Body mass index (BMI) < 14kg/m² for those over 17 years of age, BMI < 13.2kg/m² for those aged 15-16 and BMI < 12.7kg/m² for those aged 13-14.
  * Confusion
  * Bradycardia <40/min, Tachycardia
  * Blood pressure < 80/50mmHg
  * Hypothermia <35.5°C
  * Severe metabolic disorders: hypokalemia < 2.5 mmol/l, hyponatremia < 125mmol/l or hypernatremia > 150 mmol/l, hypophosphoremia < 0.5 mmol/l
  * Acetonuria, hypoglycemia < 0.6g/l
  * Creatinine elevation > 100micromol/l
  * Cytolysis > 4N
  * Leuconeutropenia <1000/mm3
  * Thrombocytopenia <6000000/mm3
  * Suicide attempt in the last month before inclusion
  * Receiving benzodiazepine treatment outside the prescription limits.
* Psychotic patients or patients with psychoactive substance addiction according to MINI KID criteria (Sheehan DV et al. Reliability and validity of the Mini International Neuropsychiatric Interview for children and adolescents (MINI Kid). J Clin Psychiatry 2010;71(3):313-326).

Ages: 13 Years to 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2021-06-20 (Actual); Primary Completion 2027-03-20 (Estimated); Study Completion 2028-09-20 (Estimated)

PRIMARY OUTCOMES:
Body Shape Questionnaire | 12 months
  The Body Shape Questionnaire (BSQ) measures concerns about body shape. The BSQ can be divided into 4 sub scores: "avoidance and social shame of body exposure", "body dissatisfaction with lower body parts", "use of laxatives and vomiting to reduce body dissatisfaction" and "inappropriate cognitions and behaviours to control weight".

SECONDARY OUTCOMES:
Eating Disorder Inventory | 12 months
  Eating Disorder Inventory (EDI-2) is a self questionnaire to assess the severity of symptoms of eating disorders and to evaluate their changes

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France